CLINICAL TRIAL: NCT02501213
Title: A Randomized Cross-over Trial Evaluating the Efficacy of Diuretics for Symptomatic Malignant Ascites Episodes in Advanced Palliative Stage of Cancer
Brief Title: Evaluation of the Efficacy of Diuretics for Symptomatic Malignant Ascites Episodes in Advanced Stage of Cancer (DIASC)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Centre Oscar Lambret (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DIASC-1507
Record Dates: First submitted 2015-07-02; First posted 2015-07-17 (Estimated); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Cancer
Keywords: Diuretic; Malignant ascites
MeSH Terms: conditions — Neoplasms | interventions — Spironolactone; Furosemide; Canrenoic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A : observation (No Intervention): Clinical monitoring and best supportive care.
- B : diuretics (Active Comparator): Diuretics (spironolactone +/- Furosemide) are administered the day after the paracentesis and until the next episode requiring paracentesis.
  Interventions: Drug: Spironolactone (+/- Furosemide)

INTERVENTIONS:
Drug: Spironolactone (+/- Furosemide) — Administration of spironolactone alone 100 mg/day each morning, increased in increments of 100 mg / week to a maximum of 400 mg / day in the absence of efficiency. In case of ineffectiveness or hyperkalemia: addition of Furosemide 40 mg / day increased in increments of 40 mg / week to a maximum of 160 mg / day in the absence of efficiency.
  Other Names: Spiroctan; Aldactone
  Arms: B : diuretics

SUMMARY:
While some authors recommend diuretics as the first treatment to initiate for symptoms caused by malignant ascites (MA), their prescription is variable. No randomized, controlled study has assessed their benefit in this context. According to literature, diuretics may bring relief in about 40% of cases, regardless of primary tumor.

The purpose of our study is to assess the effectiveness of diuretic treatment according to Serum Ascites Albumin Gradient (SAAG) measured before treatment. Judgment criteria is the time elapsed between recurrent MA that requires paracentesis. The investigators will also examine whether SAAG and serum levels of renin and aldosterone can predict symptom response to diuretics.

DETAILED DESCRIPTION:
Patients eligible for the trial and having signed their consent to participate will be randomized to arm A or B.

Treatment order is randomly attributed to patients at the 1st paracentesis, after the reception of the laboratory results necessary to evaluate SAAG value. Randomization is stratified 1:1 according to SAAG values (≥ or < to 11g/L) and Systemic treatment (yes or not)

* Patients randomized to arm A will be observed until the next episode requiring paracentesis (due to clinical symptoms : abdominal pain or heaviness, dyspnoea, orthopnoea, nausea/vomiting, anorexia, early satiety, gastro-oesophageal reflux, lower limb and genital oedema), at which time they will receive arm B (diuretics), in absence of contra-indication to diuretic treatment.
* Patients randomized to arm B will receive diuretics until the next episode requiring paracentesis, at which time they will receive arm A (observation).

Patients will have a physical assessment within 24 hours prior to the start of treatment, once every two weeks for patients randomized in arm A and each week for patients randomized in arm B, at cross-over and at the end of the study. Patient will also have a biological assessment within 24 hours prior to the start of treatment, twice a week for patients randomized in arm B, at cross-over and at the end of the study. Finally, they will address a quality of life questionnaire (QLQ-C15-PAL) prior to the start of treatment, at cross-over and at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced stage cancer
* First episode of malignant ascites
* Grade 2 or 3 ascites
* Clinically symptomatic ascites requiring paracentesis due to : abdominal pain or heaviness, dyspnoea, orthopnoea, nausea/vomiting, anorexia, early satiety, gastro-oesophageal reflux, lower limb and genital oedema
* Age ≥ 18 years
* Performance status ≤ 3
* Life expectancy ≥ 1 month
* Absence of contra-indication to diuretic treatment
* Patient regularly followed up by a palliative care or supportive care team
* Signed and dated informed consent

Exclusion Criteria:

* Hepatic disorders : cirrhosis, hepatitis, hepatocellular insufficiency, hepatic encephalopathy
* Non malignant ascites
* Hydroelectrolytic disorders: hyponatremia (< 130 mmol/L) or hyperkaliemia (> 5 mmol/L) or severe hypokaliemia (< 3 mmol/L)
* Functional acute renal insufficiency
* Urinary disorders : Obstruction in the urinary tract, Oliguria/anuria
* Chronic renal failure
* Patient unable to swallow
* Sulfamides allergy
* Hypersensitivity to spironolactone or to any of the excipients
* Hypersensitivity to furosemide or to any of the excipients
* Pregnant or breastfeeding women
* Patient under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-05-30 (Actual); Primary Completion 2017-11-23 (Actual); Study Completion 2018-12-24 (Actual)

PRIMARY OUTCOMES:
Time between symptomatic malignant ascites episodes requiring paracentesis | Patients will be followed until their third malignant ascites episode, an expected average of 30 days.

SECONDARY OUTCOMES:
Tolerance | Up to 30 days after the last administration of the product
  Adverse events and serious adverse events related to diuretic treatment according to NCI-CTCAE v4.0
Quality of life based on the EORTC (European Organization for Research and Treatment of Cancer) QLQ-C15-PAL | At baseline (prior to the start of treatment)
Quality of life based on the EORTC (European Organization for Research and Treatment of Cancer) QLQ-C15-PAL | At cross-over (approximately 15 days after inclusion)
Quality of life based on the EORTC (European Organization for Research and Treatment of Cancer) QLQ-C15-PAL | At the end of the study (up to 6 months).
Description of the patterns of prescription of diuretics | During randomization in arm B (that is to say during approximately 15 days between the first and the second or between the second and the third milgnant ascites episode).
  Growth pattern doses of diuretics, decrement pattern doses of diuretics, maintenance doses of diuretics, maximum doses reached of diuretics.
Predictive factors of response to diuretics : Serum Ascites Albumin Gradient (SAAG) | Within 24 hours prior to the start of treatment
Predictive factors of response to diuretics : renin aldosterone plasmatic level | Within 24 hours prior to the start of treatment
Predictive factors of response to diuretics : SAAG | Twice a week for patients randomized in arm B
Predictive factors of response to diuretics : renin aldosterone plasmatic level | Twice a week for patients randomized in arm B
Predictive factors of response to diuretics : SAAG | At cross-over (approximately 15 days after inclusion)
Predictive factors of response to diuretics : renin aldosterone plasmatic level | At cross-over (approximately 15 days after inclusion)
Predictive factors of response to diuretics : SAAG | At the end of the study (up to 6 months).
Predictive factors of response to diuretics : renin aldosterone plasmatic level | At the end of the study (up to 6 months).

CONTACTS AND LOCATIONS:
Overall Officials: Vincent GAMBLIN, MD, Principal Investigator — Centre Oscar Lambret
Locations (15):
- France (15):
  - Centre Hospitalier Intercommunal Compiègne-Noyon, Compiègne
  - Polyclinique de Grande Synthe, Grande-Synthe
  - CHRU Lille, Lille
  - Hôpital Saint Vincent de Paul, Lille
  - Centre Oscar Lambret, Lille
  - Institut Curie, Paris
  - Hôpital Jean Jaurès, Paris
  - GH Diaconesses Croix St Simon, Paris
  - Hôpital Lyon Sud, Pierre-Bénite
  - Institut Jean Godinot, Reims
  - Centre Eugène Marquis, Rennes
  - Centre Paul Strauss, Strasbourg
  - Centre Hospitalier Tourcoing, Tourcoing
  - Polyclinique Vauban, Valenciennes
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No